CLINICAL TRIAL: NCT04468490
Title: Adherence to Breakthrough Cancer Pain (BTcP) European Guidelines: an Observational Prospective Study.
Brief Title: Treatment of Breakthrough Cancer Pain According to European Guidelines
Acronym: BEG
Status: Terminated | Type: Observational
Why Stopped: Low enrollment rate
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Responsible Party: Sponsor
Other Study IDs: 155(A)WO19191
Record Dates: First submitted 2020-07-01; First posted 2020-07-13 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Breakthrough Cancer Pain
Keywords: Breakthrough cancer pain; Cancer; BTcP; Background pain
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP A: Patients adherent to BTcP European Guidelines
- GROUP B: Patients non Adherent to BTcP European Guidelines

SUMMARY:
Pain is a frequent symptom in cancer patients with a negative impact on the quality of life (QoL).Breakthrough cancer pain (BTcP) is defined as "a transient exacerbation of pain, manifesting spontaneously or related to a specific predictable or unpredictable triggering factor, despite stable and adequately controlled basal pain". The present study assesses the percentage of patients who are treated according to the European guidelines (ESMO, 2018) for BTcP management in 4 European countries and the impact of the adherence to guidelines on patients' pain relief and QoL.

DETAILED DESCRIPTION:
Typical BTcP episodes are of short duration (15-30 minutes/episode), moderate to severe intensity and rapid onset (maximum peak between 3-15 minutes). The best management of BTcP requires a thorough evaluation to tailor the treatment strategies. Indeed, patients with breakthrough pain should have this pain specifically assessed, starting from the appropriate diagnosis. Recently developed European guidelines support this approach and recommend treating BTcP using rapid-onset opioids (ROOs), with pharmacodynamics that mirror the quick start and short duration of the pain episode.Nevertheless, despite the drug treatment for BTcP has undergone knowledge advances in recent years and several guidelines have been published, this condition is still often inadequately managed.

The present study will assess the percentage of patients who are treated according to the European guidelines for BTcP management in 4 European countries and the impact of the adherence to guidelines on patients' pain relief and QoL.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any ethnic origin of ≥ 18 years.
* Patients diagnosed with locally advanced or recurrent metastatic cancer (histologic or cytologic diagnosis), with BTcP, as assessed by the Investigator.
* Opioid-tolerant patients receiving doses of oral morphine equivalent daily doses (OMEDD) of at least 60 mg.
* Drugs for BTcP treatment, if any, must be used according to the relevant SmPC.
* Eastern Cooperative Oncology Group (ECOG) performance status with a score of 0, or 1, or 2.
* Patients with life expectancy > 3 months.
* Patients legally capable of giving their consent to participate in the study and available to sign and date the written informed consent.

Exclusion Criteria:

* Patients with previous or current history of a clinically significant neurological/psychiatric disorder and/or any substance abuse or dependence that, according to the Investigator's judgement, can impair the study end-points/results.
* Patients who have been taking antidepressants and/or drugs acting on pain and who take them on a regular basis during the observation period, can be enrolled.
* Any medical condition or situation complicating the collection of study data, as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with BTcP.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients treated according to 2018 ESMO European Guideline guidelines for BTcP. | 4 weeks of observation
  Percentage of BTcP treatment guideline adherent vs non-adherent patients, in the 4 weeks of observation (V2)

SECONDARY OUTCOMES:
APM algorithm | 0, 1, 2, 3, 4 weeks of observation
  BTcP diagnosis by APM algorithm observation (V0, telephone contact1, V1, telephone contact2, V2)
Tool-BAT | at 0, 1, 2, 3, 4 weeks of observation
  BTcP assessment by Tool-BAT (V0, telephone contact1, V1, telephone contact2, V2)
EORTC QLQ-C30 | at 0, 1, 2, 3, 4 weeks of observation
  Quality of life assessed by the questionnaire EORTC: 28 questions from 1 to 4 (there are not wrong or right answers) + 2 questions from 7 point scales from 1 (very poor) to 7 (excellent)
Patient Global Impression of Change (PGIC) | at 0, 2 and 4 weeks of observation
  Global impression of clinical condition assessed by the Patient through 7 point scales from 1 (very much improved) to 7 (very much worse).
Healthcare resources consumed due to cancer pain (Number of specialist/GP visits) | at 2 and 4 weeks of observation
  Number of specialist/GP visits due to cancer pain during the observation period
Healthcare resources consumed due to cancer pain (Number of hospitalizations) | at 2 and 4 weeks of observation
  Number of hospitalizations due to cancer pain during the observation period
Healthcare resources consumed due to cancer pain (Length of hospitalizations) | at 2 and 4 weeks of observation
  Length of hospitalizations (days) due to cancer pain during the observation period
Healthcare resources consumed due to cancer pain (Number of admittances to ER) due to cancer pain) | at 2 and 4 weeks of observation
  Number of admittances to ER due to cancer pain during the observation period

CONTACTS AND LOCATIONS:
Locations (1):
- Nzoz Zespół Medyczno Opiekuńczy Alicja Kluczna, Dąbrowa Górnicza, Poland

IPD SHARING:
Plan to Share IPD: No